CLINICAL TRIAL: NCT07174882
Title: Evaluation of the Clinical Course of Non-erosive Reflux Disease and Assessment of the Esophageal Mucosa Resistance Before and After Complex Therapy
Brief Title: Evaluation of the Clinical Course of NERD and Assessment of the Esophageal Mucosa Resistance
Status: Active, not recruiting | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 29091973
Record Dates: First submitted 2024-12-02; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2024-12

CONDITIONS: Non-Erosive Gastro-Esophageal Reflux Disease; Gastroesophageal Reflux Disease (GERD)
Keywords: GERD; NERD; rebamipide; epithelial resistance; cytoprotection
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main group (intervention group): 30 patients: Participants in the main group will receive combination therapy with a proton pump inhibitor and rebamipide for 4 weeks.
- Control group: 30 patients: Participants in the control group will receive monotherapy with a proton pump inhibitor for 4 weeks.

SUMMARY:
GERD is characterized by a high prevalence (about 13.3%) and is associated with a deterioration in the quality of life, as well as an increased risk of esophageal adenocarcinoma and a rise in the number of refractory cases. NERD is one of the forms of GERD, accounting for about 70% of all cases, and is characterized by symptoms that reduce the quality of life. Although proton pump inhibitors (PPIs) are the basic therapy for NERD, up to 40% of patients do not achieve an optimal clinical outcome. GERD symptoms seriously affect the quality of life and performance, which makes the study of complex therapy relevant. One of the mechanisms of GERD is a violation of the barrier function of the esophageal mucosa, associated with an increase in epithelial permeability due to the dysfunction of intercellular junction proteins, such as claudins and occludin. The study of methods to increase tissue resistance and cytoprotection, together with acid-suppressive therapy, is a promising direction, especially for refractory forms of NERD. It is relevant to study the complex treatment of NERD in order to change the clinical course of the disease and improve the tissue resistance of the esophageal mucosa. These hypotheses and theses emphasize the need for a comprehensive approach to the treatment of NERD and a research focus on improving the barrier functions of the esophagus

DETAILED DESCRIPTION:
The relevance of gastroesophageal reflux disease (GERD) in clinical practice today is associated with its high prevalence, significant reduction in patients' quality of life, increased risk of esophageal adenocarcinoma, and a growing number of cases resistant to standard antisecretory therapy. Recent estimates indicate a global prevalence of GERD at approximately 13.3%. Non-erosive reflux disease (NERD) is a GERD phenotype characterized by reflux-induced symptoms that impair quality of life without esophageal mucosal erosions detectable by conventional endoscopy, and occurring in the absence of ongoing antisecretory therapy. According to the literature, about 70% of GERD cases are attributed to the NERD. Proton pump inhibitors (PPIs) are the cornerstone of NERD therapy; however, studies reveal that up to 40% of patients do not achieve optimal clinical outcomes with PPI therapy. Notably, the significant impact of GERD symptoms on patients' quality of life and work capacity represents a crucial medical and social issue, underscoring the relevance of exploring combination therapies and addressing the key pathogenetic factors of the disease.

One of the leading mechanisms in the development of the disease is the impaired barrier function of the esophageal mucosa, a critical aspect of which is increased epithelial permeability due to disrupted intercellular resistance resulting from the dysfunction of tight junction proteins. Major proteins involved in intercellular adhesion include claudin-1, claudin-3, claudin-4, and occludin, whose primary cytoprotective role is to prevent the diffusion of H+ ions and other active luminal substances into the esophageal mucosa. Investigating ways to enhance tissue resistance and cytoprotection by targeting the barrier function of the esophageal mucosa, alongside standard acid-suppressive therapy, represents a promising approach in NERD treatment, particularly for refractory cases.

Thus, it is pertinent to study the role of comprehensive treatment of NERD in altering the clinical course of the disease and the tissue resistance parameters of the esophageal mucosa.

2. Novelty of the Proposed Topic Based on Literature Sources and Patent Documentation

The novelty of this study lies in the comprehensive examination of the following parameters:

1. The impact of combination therapy on the clinical and morphological characteristics of NERD.
2. The influence of combination therapy on the expression of intercellular adhesion proteins of the esophageal mucosa.
3. The relationship between tissue resistance parameters of the esophageal mucosa, motor function efficacy, inflammation severity, and the occurrence of symptoms characteristic of NERD.
4. Evaluation of daily pH-impedance metrics, including esophageal mucosa impedance through the baseline impedance level measurements, before and after combination therapy.
5. Assessment of high-resolution manometry parameters before and after the application of combination therapy.

Research Aim: The aim of this study is to enhance the effectiveness of treating non-erosive reflux disease (NERD) patients by implementing a novel therapeutic approach aimed at achieving a complete clinical response and improving the tissue resistance of the esophageal mucosa.

Research Objectives:

1. Evaluate the impact of combination therapy with Rebamipide and a proton pump inhibitor (PPI) on the clinical course of NERD after four weeks of treatment compared to PPI monotherapy. Assess the intensity of symptoms using a Likert scale questionnaire (including intensity of heartburn, regurgitation, chest pain, belching, cough, and sensation of mucus in the throat) before treatment and 4 weeks after the start of therapy.
2. Compare the laboratory and instrumental characteristics of NERD patients before and after combination therapy with PPI and Rebamipide:

   2.1 Assess 24-hour pH-impedance measurements, including acid exposure time, gastroesophageal refluxes number, DeMeester index, reflux type, reflux pattern, symptom index (SI), symptom association probability (SAP), mean nocturnal basal impedance (MNBI) before therapy and 4 weeks after the start of therapy.

   2.2 Study high-resolution manometry measurements with assessment of the following parameters: distal contractile integral, lower esophageal sphincter pressure, transient LES relaxations, esophagogastric junction complex type
3. Evaluate inflammatory changes in the esophageal mucosa based on data from esophagogastroduodenoscopy (EGD) before and after combination therapy.
4. Examine the inflammatory changes in the esophageal mucosa (such as dilated intercellular spaces, intraepithelial eosinophils, intraepithelial neutrophils, intraepithelial mononuclear cells, basal cell hyperplasia, elongation of papillae in the lamina propria, and spongiosis) through morphological examination before treatment and again 4 weeks after the start of therapy. Assess intercellular space width through morphometry.
5. Analyze the effect of combination therapy on enhancing tissue resistance of the esophageal mucosa by influencing the expression of intercellular adhesion proteins the (claudin 1, claudin 3, claudin 4, and occludin) by immunohistochemistry both before treatment and 4 weeks after the start of therapy.
6. Assess the safety of combination therapy with Rebamipide and PPI in the treatment of NERD patients.

Study Design:

An open-label, prospective, randomized, single-center clinical study.

Study Subjects and Planned Sample Size Justification:

The study will include 60 patients diagnosed with NERD who meet the inclusion criteria and do not have any exclusion criteria.

Evaluated Outcomes (Primary and Secondary Endpoints):

Primary Endpoints (Direct Outcomes): Assessment of the severity of symptoms characteristic of NERD, evaluation of inflammatory changes in the esophageal mucosa based on morphological study data, and assessment of the expression of tight junction markers using immunohistochemistry four weeks after the start of therapy.

Secondary Endpoints (Indirect Outcomes): Evaluation of pH-impedance metrics, including mucosal impedance of the esophagus, and high-resolution manometry three weeks after the start of therapy.

Planned Research Methods (Statistical Analysis Techniques):

The study involves analyzing clinical, anamnestic, and laboratory-instrumental data in 60 NERD patients before and after combination therapy:

Collection of anamnesis and assessment of the objective status Completion of a Likert scale questionnaire (intensity of heartburn, regurgitation, retrosternal pain, belching, cough, mucus formation in the larynx) Clinical examination (complete blood count, general urine analysis, biochemical blood analysis); ECG with 12 leads EGD with biopsy sampling from the lower third of the esophageal mucosa, morphological study with assessment of inflammatory mucosal changes and intercellular space width Investigation of esophageal mucosa tight junction markers: claudin-1, claudin-3, claudin-4, occludin via immunohistochemistry (IHC) 24-hour pH-impedance monitoring High-resolution esophageal manometry

Anticipated Research Outcome:

The research aims to determine the effectiveness of combination therapy in the clinical course of NERD and explore its impact on the tissue resistance of the esophageal mucosa in comparison with the standard PPI monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. The availability of written informed consent from the patient to participate in the study.
2. Patients aged over 18 years.
3. Gender: both men and women.
4. The patient must be able to independently fill out questionnaires and assess their condition using scales.
5. A confirmed diagnosis of non-erosive reflux disease.

Exclusion Criteria:

1. The voluntary withdrawal of consent to participate in the study by the patient.
2. Pregnancy.
3. The patient experienced a serious adverse event, the relationship of which to the study drug is classified as definite, probable, or possible.
4. The patient is receiving/requires additional treatment that may affect the efficacy parameters being studied.
5. Protocol violations that, in the opinion of the investigator, are significant for the results of the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient both gender from 18 to 75 years old
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-12-13 (Estimated)

PRIMARY OUTCOMES:
Assess the intensity of symptoms | Before treatment and 4 weeks after the start of therapy
  Assess the intensity of symptoms using a SYMPTOM INTENSITY QUESTIONNAIRE ON THE LIKERT SCALE (including intensity of heartburn, regurgitation, chest pain, belching, cough, and sensation of mucus in the throat).
  5-point scale:
  1. Symptom absent
  2. Mild symptom, occasionally present
  3. Moderate symptom
  4. Severe symptom
  5. Persistent symptom
Examine the inflammatory changes in the esophageal mucosa. | Before treatment and again 4 weeks after the start of therapy.
  Examine the inflammatory changes in the esophageal mucosa (such as dilated intercellular spaces, intraepithelial eosinophils, intraepithelial neutrophils, intraepithelial mononuclear cells, basal cell hyperplasia, elongation of papillae in the lamina propria, and spongiosis) through morphological examination.
Study the expression of tight junction proteins in esophageal mucosa. | Before treatment and 4 weeks after the start of therapy.
  Study the expression of tight junction proteins in esophageal mucosa samples by immunohistochemistry.

SECONDARY OUTCOMES:
Assess the сhange in Acid Exposure Time (%) | Before treatment and 4 weeks after the start of therapy
  Metric defining abnormal esophageal acid burden, measured by 24-hour pH-impedance monitoring.
Change in Total Number of Gastroesophageal Reflux Episodes | Before treatment and 4 weeks after the start of therapy
  The total number of reflux episodes (including acidic, slightly acidic, and slightly alkaline), measured by 24-hour pH-impedance monitoring.
Change in Number of Proximal Reflux Episodes | Before treatment and 4 weeks after the start of therapy
  The number of reflux episodes reaching 17 cm above the lower esophageal sphincter, measured by 24-hour pH-impedance monitoring.
Change in Composition of Reflux Episodes (Liquid, Mixed, Gas) | Before treatment and 4 weeks after the start of therapy
  The number of reflux episodes categorized by their composition (liquid, mixed, gas), measured by 24-hour pH-impedance monitoring.
Change in Mean Nocturnal Baseline Impedance (MNBI) (Ohms) | Before treatment and 4 weeks after the start of therapy
  An indicator evaluating esophageal mucosal integrity, measured by 24-hour pH-impedance monitoring.
Change in Lower Esophageal Sphincter Pressure (mmHg) | Before treatment and 4 weeks after the start of therapy
  Metric to assess the barrier function of the esophagus, measured by high-resolution manometry.
Change in Distal Esophageal Contractile Integral (mmHg · cm · sec) | Before treatment and 4 weeks after the start of therapy
  Metric to assess the strength of esophageal peristalsis (esophageal muscle contraction), measured by high-resolution manometry.
Change in Number of Transient Lower Esophageal Sphincter Relaxations (TLESRs) | Before treatment and 4 weeks after the start of therapy
  The number of spontaneous lower esophageal sphincter relaxations not triggered by swallowing, which are a primary cause of gastroesophageal reflux, measured by high-resolution manometry.

CONTACTS AND LOCATIONS:
Locations (1):
- V.Kh.Vasilenko Clinic of Propedeutics of Internal Diseases, Gastroenterology and Hepatology, I.M.Sechenov First Moscow State Medical University (Sechenov University). Gastroenterology department, outpatient clinic., Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided